CLINICAL TRIAL: NCT00094432
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of Aripiprazole in the Treatment of Patients With Bipolar I Disorder With a Major Depressive Episode. CN138-146 LT is the 26-week Open Label Extension Phase of the Above Titled Protocol, CN138-146 ST.
Brief Title: A Study of Aripiprazole in Patients With Bipolar I Disorder With a Major Depressive Episode
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN138-146
Record Dates: First submitted 2004-10-18; First posted 2004-10-19 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2008-06

CONDITIONS: Bipolar I Disorder
Keywords: depressed
MeSH Terms: conditions — Consciousness Disorders | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A1 (Active Comparator)
  Interventions: Drug: Aripiprazole
- A2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole — Tablets, Oral, 10mg (2 5mg tablets), Once daily, 8 weeks.
  Other Names: Abilify
  Arms: A1
Drug: Placebo — Tablets, Oral, 0 mg, Once daily, 8 weeks.
  Arms: A2

SUMMARY:
The purpose of this study is to evaluate several doses of aripiprazole in patients with bipolar depression.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18-65
* Have experienced a prior manic episode that required treatment with a mood stabilizer or antipsychotic, and now meet criteria for a major depressive episode.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650
Dates: Start 2004-06; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline to endpoint on the MADRS total score.

SECONDARY OUTCOMES:
Clinical Global Impression - Bipolar Version
Severity of illness score depression
Mean change from baseline to endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (40):
- United States (40):
  - Local Institution, Mesa, Arizona
  - Local Institution, La Mesa, California
  - Local Institution, La Palma, California
  - Local Institution, Long Beach, California
  - Local Institution, Redlands, California
  - Local Institution, San Diego, California
  - Local Institution, Sherman Oaks, California
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Coral Springs, Florida
  - Local Institution, Jacksonville, Florida
  - Local Institution, St. Petersburg, Florida
  - Local Institution, Marietta, Georgia
  - Local Institution, Edwardsville, Illinois
  - Local Institution, Oak Brook, Illinois
  - Local Institution, Springfield, Illinois
  - Local Institution, Lafayette, Indiana
  - Local Institution, Newton, Kansas
  - Local Institution, New Orleans, Louisiana
  - Local Institution, Shreveport, Louisiana
  - Local Institution, Baltimore, Maryland
  - Local Institution, St Louis, Missouri
  - Local Institution, Clementon, New Jersey
  - Local Institution, Albuquerque, New Mexico
  - Local Institution, Brooklyn, New York
  - Local Institution, Elmsford, New York
  - Local Institution, New York, New York
  - Local Institution, Raleigh, North Carolina
  - Local Institution, Dayton, Ohio
  - Local Institution, Media, Pennsylvania
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, Columbia, South Carolina
  - Local Institution, DeSoto, Texas
  - Local Institution, Houston, Texas
  - Local Institution, Wichita Falls, Texas
  - Local Institution, Salt Lake City, Utah
  - Local Institution, Charlottesville, Virginia
  - Local Institution, Midlothian, Virginia
  - Local Institution, Bellevue, Washington
  - Local Institution, Charleston, West Virginia